CLINICAL TRIAL: NCT05578027
Title: Change in Skin Surface Temperature at the Knee Area on Both Sides When Using Mild Moxibustion Manipulation at Mingmen Acupoint With Moxa Stick: A Pilot Study
Brief Title: Change in Skin Surface Temperature at the Knee Area on Both Sides When Using Mild Moxibustion Manipulation at Mingmen Acupoint With Moxa Stick
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bui Pham Minh Man (Other)
Responsible Party: Sponsor-Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 677/HDDD-DHYD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Moxibustion; Skin surface temperature

STUDY DESIGN:
Intervention Model Description: A pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: P1M2 (Experimental): 19 participants received mild moxibustion manipulation at the control acupoint (the left side Pishu acupoint) and the research acupoint (Mingmen) in the first and the second trial phase, respectively. In each trial phase, skin surface temperature at the local stimulated area and the knee area on both sides will be recorded.
  Interventions: Procedure: Mild moxibustion with moxa stick
- Group B: M1P2 (Experimental): 19 participants received mild moxibustion manipulation at the research acupoint (Mingmen) and the control acupoint (the left side Pishu acupoint) in the first and the second trial phase, respectively. In each trial phase, skin surface temperature at the local stimulated area and the knee area on both sides will be recorded.
  Interventions: Procedure: Mild moxibustion with moxa stick

INTERVENTIONS:
Procedure: Mild moxibustion with moxa stick — To conduct this intervention, we used moxa sticks which were 1.5 cm in diameter, 13 cm long, and weighed 12 gram to perform mild moxibustion manipulation at the control acupoint (the left side Pishu acupoint) or Mingmen acupoint in 2 trial phases. The main ingredient of the moxa was dried mugwort leaf, produced in Vietnam. All moxa materials were obtained from the Sai Gon TCS Co., Ho Chi Minh City, Vietnam.

SUMMARY:
Moxibustion plays an important role in Traditional Medicine treatments, which treats and prevents diseases by burning a herb preparation containing Moxa (Artemisia vulgaris, Mugwort) to stimulate the meridians of human body. Moxibustion is considered a safe and effective traditional therapy. Mild moxibustion is a kind of therapeutic method which characterized by wide indications, simple manipulation and comfortable feeling, is commonly used in clinical treatment. Mingmen acupoint located on the midline of the lower back, in the depression below the spinous process of the 2nd lumbar vertebra (L2). Its indications include Yang-deficiency syndrome, Cold-Stagnation syndrome, Cold Excessive syndrome,... and it is closely related to the knee area through the path of Thoroughfare Vessel (one of the Eight Extraordinary Vessels). In our study, we investigate the change in skin surface temperature at the knee area on both sides when using mild moxibustion manipulation at Mingmen acupoint with moxa stick in healthy volunteers.

DETAILED DESCRIPTION:
Participants and Methods: A randomized controlled trial is conducted by comparing the change in skin surface temperature before and after using mild moxibustion manipulation at the research acupoint (Mingmen (GV-4) acupoint) or the control acupoint (the left side Pishu (BL-20) acupoint) in healthy volunteers. A total of 38 participants will undergo 2 trial phases, corresponding to 2 times of moxibustion in 8 days, each time is 7 days apart. In the first trial phase: participants received moxibustion at left side Pishu (BL-20) acupoint. In the second trial phase: participants received moxibustion at Mingmen (GV-4) acupoint. The primary outcome was the change in skin surface temperature at the local stimulated area and the knee area on both sides when using mild moxibustion manipulation at Mingmen acupoint. This trial will be performed as a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females were individual age between enough 18 and 30 years old.
* BMI: 18.5 - 23 kg/m2
* Mental alertness, good contact, cooperation with researchers.
* Had no psychiatric stress problem during moxibustion day (confirmed by answering the DASS 21 questionaire with stress point less than 15 points).
* Had no history of cardio-vascular disease, diabetes, hyperthyroidism, hypothyroidism.
* Vital sign within normal limits:

  * Heart rates from from 60 to 99 beats/minute.
  * Systolic blood pressure between 90 and 139 mmHg.
  * Diastolic blood pressure between 60 and 89 mmHg.
  * Breathing rate: 16 ± 3 times/minute.
  * Body temperature: 36.59 ± 0.43 ℃.
  * SpO2 from 95 to 100%.
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials.
* Not currently participating in other intervention studies.

Exclusion Criteria:

* Having an inflammatory injury in the site of the skin to be investigated.
* Medical history of asthma or allergy with moxa smoke.
* Using heat therapy, for example massage, cupping therapy, acupuncture in the site of the skin to be investigated within 24 hours.
* Applying chemical or pharmaceutical products to the site of the skin to be survey before conducting the study.
* Other diseases that could affect or interfere with outcomes, including common cold or flu.
* Playing sport 2 hours before the study.
* Taking stimulants such as beer, alcohol, coffee and tobacco within 24 hours before conducting the study.
* Skin surface temperature disorders or sensation disorders at lower-back or knee area.
* Staying up at night or having insomnia before moxibustion day.
* Women during menstruation period, pregnancy, or breastfeeding.
* Currently using certain drugs which dilate blood vessels and drop in blood pressure.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in skin surface temperature at the local stimulated area when using mild moxibustion manipulation at Mingmen acupoint | During procedure
Change in skin surface temperature at the knee area on both sides when using mild moxibustion manipulation at Mingmen acupoint | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: Deng H, Shen X. The mechanism of moxibustion: ancient theory and modern research. Journal of Evidence-Based Complementary and Alternative Medicine. 2013;2013 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3789413/
- See also: Sun C, Li Y, Kuang J, Liang X, Wu J, Ji C. The thermal performance of biological tissue under moxibustion therapy. Journal of thermal biology. 2019;83:103-111. — https://pubmed.ncbi.nlm.nih.gov/31331508/
- See also: Coiffard B, Diallo AB, Mezouar S, Leone M, Mege JL. A Tangled Threesome: Circadian Rhythm, Body Temperature Variations, and the Immune System. Biology (Basel). Jan 18 2021;10(1)doi:10.3390/biology10010065 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7829919/
- See also: Yang Y, Ji L, Li G, Deng X, Cai P, Guan LJJoTCM. Differences in thermal effects of moxibustion at Zusanli (ST 36) and Hegu (LI 4) on various facial areas in healthy people. 2012;32(3):397-403. — https://pubmed.ncbi.nlm.nih.gov/23297563/